CLINICAL TRIAL: NCT02840942
Title: Socially Assistive Robots to Reduce Children's Pain During Peripheral IV Placement
Brief Title: Robots to Reduce Pain During IV Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Margaret Trost MD, Attending Physician, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-14-00231
Record Dates: First submitted 2016-05-20; First posted 2016-07-21 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Pain; Anxiety
Keywords: intravenous line; robot
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-robot (No Intervention): Patients will interact with Child Life as per usual routine, no robot condition
- Coping Robot (Experimental): Robot will play coping game with children. Robot will speak and child will respond by touching tablet. Child life still present.
  Interventions: Behavioral: Coping Robot
- Non-coping Robot (Experimental): Robot will play distraction only game, in addition to Child Life and routine cares
  Interventions: Behavioral: Non-coping Robot

INTERVENTIONS:
Behavioral: Coping Robot — Socially assistive robot "MAKI" will interact with children via tablet game designed to teach coping skills.
  Arms: Coping Robot
Behavioral: Non-coping Robot — Socially assistive robot "MAKI" will interact with children via tablet game designed to be distraction only.
  Arms: Non-coping Robot

SUMMARY:
Peripheral intravenous catheters (IVs) are utilized in the majority of hospitalized children. The placement of IVs requires significant staff time, contributes to health care costs, and causes pain and distress in the patients receiving them. Techniques currently used at Children's Hospital Los Angeles (CHLA) to reduce children's anxiety and increase success of IV placement center depends on members of the Child Life Department distracting patients during insertion. Recent literature has suggested that humanoid robots can be a powerful form of distraction and lead to decreased pain during painful procedures in children. Work done by the University of Southern California (USC) Interaction Lab has shown that socially assistive robots can use techniques more complex than pure distraction to lead to a human-robot interaction that is perceived as more positive by the human. The investigators propose a project pairing children receiving an IV with either a (1) Child Life staff member only (2) pure distraction robot + Child Life or (3) an robot teaching coping skills + Child Life with a goal of reduced pain. Pain will be measured by participant self-report, family member perceived pain, parasympathetic activation, and pain behaviors as measured by video.

DETAILED DESCRIPTION:
At USC University Park, computer science collaborators have programmed the robot to speak the script which will be used for interaction with participants (see additional supporting documents).

At CHLA, patients arriving to the radiology suite for IV placement prior to MRI and utilizing Child Life Services will be approached and consented for inclusion. No participant will receive a IV purely for the purpose of the study; only participants already ordered to receive IV by the medical team will be included. After consent participants will be randomized in blocks using a random-condition generating document to one of three test conditions: (1) control, with the usual distraction services provided by one of the hospital's child life specialists (2) usual child life + non-coping robot or (2) usual child life + coping robot.

Prior to the procedure participant's parent (or legal guardian) will complete a short survey related to pain with previous IV insertions, anxiety related to procedures, and attitudes toward robots. Participant's parent/guardian will also complete a validated measure of child temperament. Participants will complete a baseline measure of their temperament. Participants will then rate current level of pain using the Wong-Baker FACES scale. Participant's anxiety level will be assessed using the Children's Fear Scale. Participant's baseline heart rate and blood pressure is recorded.

The IV placement itself will be video recorded for all conditions. Independent assessors not aware of the research aims will review the tape to score measures of the strength of robot-child interaction and pain behaviors. One research team member will record the number of attempts needed to place the IV. A trained research team member will be responsible for operating the robot if randomized to that condition.

The robot used is the MAKI - an open-source 3D printable robot designed by Hello Robo Inc. The company has not provided any funding to this project. During the interaction the robot will speak in a child-like, gender neutral voice. It will ask short questions of participants and have pre-recorded response options (see MAKI script in supporting documents). Participants will interact with either child life or the robot by touching tablets. This is a minimum risk study, similar to the risk involved in watching a video on a screen. The robot is small and only moves its facial features, participants are not touching it.

Pre- and post-intervention participants will repeat the FACES and Fear Scales. The participant and parent/guardian will then be given a short post-survey regarding thoughts on the utility of the interaction and the amount of the participant's pain. Heart rate will be monitored continuously throughout the interaction. Videos will be evaluated using the modified Yale Preoperative Anxiety Index and The Child-Adult Medical Procedure Interaction Scale-Short Form (CAMPIS-SF).

ELIGIBILITY:
Inclusion Criteria:

* Speaks English or Spanish
* Age limits
* would be getting IV and child life regardless of participation in study

Exclusion Criteria:

* severe developmental delay (parent assessment)
* afraid of robots

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Change in Pain Scale Score from baseline to post-intervention | through study completion, an average of 1 hour
  Using Wong-baker faces pain scale

SECONDARY OUTCOMES:
IV placement attempts | through study completion, an average of 1 hour
  record raw number of attempts to compare average between arms
Patient/Child satisfaction with robot interaction | Day 1
  by survey
CAMPIS score | Day 1
  on video review
mYPAS score | Day 1
  on video review
Change in Anxiety Scale Score from baseline to post-intervention | through study completion, an average of 1 hour
  using fear faces scale
heart rate | through study completion, an average of 1 hour
  using pulse oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okita SY. Self-other's perspective taking: the use of therapeutic robot companions as social agents for reducing pain and anxiety in pediatric patients. Cyberpsychol Behav Soc Netw. 2013 Jun;16(6):436-41. doi: 10.1089/cyber.2012.0513. Epub 2013 Mar 18. PMID 23505968
- [Background] Beran TN, Ramirez-Serrano A, Vanderkooi OG, Kuhn S. Reducing children's pain and distress towards flu vaccinations: a novel and effective application of humanoid robotics. Vaccine. 2013 Jun 7;31(25):2772-7. doi: 10.1016/j.vaccine.2013.03.056. Epub 2013 Apr 24. PMID 23623861
- [Derived] Trost MJ, Chrysilla G, Gold JI, Mataric M. Socially-Assistive Robots Using Empathy to Reduce Pain and Distress during Peripheral IV Placement in Children. Pain Res Manag. 2020 Apr 9;2020:7935215. doi: 10.1155/2020/7935215. eCollection 2020. PMID 32351642